CLINICAL TRIAL: NCT01965106
Title: Phase IIA Double-Masked Randomized Sham-Controlled Trial of QPI-1007 Delivered by a Single Intravitreal Injection to Subjects With Acute Primary Angle-Closure Glaucoma (APACG)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Quark Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: QRK208
Record Dates: First submitted 2013-09-11; First posted 2013-10-18 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Glaucoma, Angle-closure, Primary, Acute
Keywords: Glaucoma, Angle-Closure; Glaucoma, Closed-Angle; Primary angle closure; Acute angle closure; Acute angle-closure glaucoma
MeSH Terms: conditions — Glaucoma; Glaucoma, Angle-Closure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- QPI-1007 Injection (Active Comparator): single intravitreal (IVT) injection of QPI-1007
  Interventions: Drug: QPI-1007 Injection
- Control (Sham Comparator): Placebo (Sham injection procedure)
  Interventions: Drug: (including placebo)

INTERVENTIONS:
Drug: QPI-1007 Injection — 1.5 mg QPI-1007 Injection
  Arms: QPI-1007 Injection
Drug: (including placebo) — Sham injection procedure
  Arms: Control

SUMMARY:
This study will assess any side effects that may occur when QPI-1007 is injected into the eye in subjects with acute primary angle-closure glaucoma, as well as how long it takes for the body to clear the drug. This study will also test whether QPI-1007, injected into the eye, helps prevent both structural damage of the nerve tissue in the eye and the loss of visual function in subjects with acute primary angle-closure glaucoma.

DETAILED DESCRIPTION:
This is a Phase IIa double-masked, single dose, randomized, sham-controlled study evaluating the safety and tolerability, and pharmacokinetics of QPI-1007 versus Control (sham procedure) in subjects with an acute attack of primary angle-closure glaucoma.

Subjects will be randomized at a ratio of 1:1 into one of two study arms: 1.5 QPI-1007 arm or Control arm (sham procedure). The study will enroll approximately 30 subjects into each arm. Randomization will be stratified by time from symptom onset to the study drug administration or sham procedure (≤72 hours and >72 hours).

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged at least 40 years or older.
* Onset of symptoms of an acute attack of primary angle-closure in the study eye within the 120 hours prior to the planned study drug administration.
* Best-corrected visual acuity (BCVA) 20/40 or better in the study eye after resolution of the acute attack.
* Received successful treatment for the acute attack of angle-closure, and have undergone laser iridotomy with intraocular pressure in the study eye <25mm Hg.
* Sufficiently clear ocular media and adequate pupil dilation to allow the optic nerve and fovea to be visualized and assessed in the study eye.
* Female subjects must be: (1) post menopausal, (2) surgically sterile, or (3) using an effective means of contraception.

Exclusion Criteria:

* Previously diagnosed with glaucoma in either eye.
* The time planned for study drug administration is more than 120 hours from the onset of the symptoms.
* History of chronic angle-closure in either eye.
* Secondary angle-closure/secondary angle-closure glaucoma in the study eye.
* Monocular subjects.
* Prior incisional intraocular surgery.
* Inability to perform a reliable visual field test on Day 0 in the study eye.
* History of panretinal photocoagulation or macular laser photocoagulation in the study eye.
* History of active malignancy within the last 5 years (however, non facial, basal cell carcinoma is allowed).
* History of myocardial infarction within the last 6 months.
* Received any drugs known to cause optic nerve or retinal toxicity within 14 days prior to dosing.
* Women who are pregnant or lactating.
* Participating in a concurrent interventional study with the last intervention occurring within 30 days prior to planned dosing with QPI-1007.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-12; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of a single intravitreal (IVT) dose of QPI-1007 as assessed by adverse events (AE) | Day 0 (after injection) through Month 4. Systemic serious AEs (SAEs) assessed as related to study drug and all ocular SAEs Month 4 to Month 6 after injection
Safety and tolerability of a single IVT dose of QPI-1007 as assessed by laboratory evaluations | Screening, Day 1, and Month 4 after injection
Safety and tolerability of a single IVT dose of QPI-1007 as assessed by vital signs and weight | Weight: Screening and Month 4; Vital signs: Screening, Days 0 (before injection), 1 and 7, and Month 4 to 6
Safety and tolerability of a single IVT dose of QPI-1007 as assessed by ophthalmic evaluations, Best Corrected Visual Acuity (BCVA) using Early Treatment Diabetic Retinopathy Study (EDTRS) chart and slit lamp exams (anterior & posterior segment) | Screening, Days 0, 1 and 7, and Month 1 to 6
Safety and tolerability of a single IVT dose of QPI-1007 as assessed by ophthalmic evaluations, Visual Field (VF) and Spectral Domain Optical Coherence Tomography (SD-OCT) | Days 0 and 7, and Month 1 to 6
Safety and tolerability of a single IVT dose of QPI-1007 as assessed by ophthalmic evaluation intraocular pressure (IOP) | Screening, Days 0 (before injection, both eyes; after injection study eye only), 1 and 7, and Month 1 to 6
Safety and tolerability of a single IVT dose of QPI-1007 as assessed by ophthalmic evaluation, Fundus Photographs (FP) | Days 0 and 7, and Month 4
Safety and tolerability of a single IVT dose of QPI-1007 as assessed by ophthalmic evaluations optic nerve head stereo photographs and contrast sensitivity | Days 0 and 7, and Month 4 and 6
Safety and tolerability of a single IVT dose of QPI-1007 as assessed by use of concomitant treatments | Days 0, 1 and 7, and Month 1 to 6

SECONDARY OUTCOMES:
QPI-1007 pharmacokinetics (PK) parameters as assessed by the peak plasma concentration (Cmax) | Pre-injection, 1, 4 and 24 hours after injection, and 7 days after injection
QPI-1007 pharmacokinetics (PK) parameters as assessed by the time to peak plasma concentration (Tmax) | Pre-injection, 1, 4 and 24 hours after injection, and 7 days after injection
Difference between QPI-1007 and control group (sham) as assessed by the prevalence of the abnormal visual fields | 4 months after injection
Difference between QPI-1007 and control group (sham) as assessed by change in the mean deviation compared to baseline | 4 months after injection
Difference between QPI-1007 and control group (sham) as assessed by progression of the visual fields compared to baseline | 4 months after injection
Difference between QPI-1007 and control group (sham) as assessed by change in the mean BCVA using the EDTRS chart compared to baseline | 4 months after injection
Difference between QPI-1007 and control group (sham) as assessed by SD-OCT parameters | 4 months after injection
Difference between QPI-1007 and control group (sham) as assessed by change in the mean contrast sensitivity compared to baseline | 4 months after injection

CONTACTS AND LOCATIONS:
Overall Officials: Avner Ingerman, M.D., MSc., Study Chair — Quark Pharmaceuticals
Locations (8):
- United States (4):
  - The Gavin Herbert Eye Institute, UC Irvine, Orange, California
  - Doheny Eye Center, UCLA, Pasadena, California
  - Robert Cizik Eye Clinic - Clinical Trials Unit, Houston, Texas
  - Dept. of Ophthalmology, University of Washington Medical Center, Seattle, Washington
- Singapore National Eye Centre, Singapore, Singapore
- Vietnam (3):
  - Hanoi Eye Hospital, Hà Nội
  - Vietnam National Institute of Ophthalmology, Hà Nội
  - Ho Chi Minh City Eye Hospital, Ho Chi Minh City